CLINICAL TRIAL: NCT03959735
Title: "Is the Use of High Intensity Interval Training (HIIT) Feasible and Acceptable Amongst Inpatients With Severe Mental Illness (SMI)?" A Pilot Study
Brief Title: High Intensity Interval Training in Severe Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRAS263996
Record Dates: First submitted 2019-05-17; First posted 2019-05-22 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2020-09

CONDITIONS: Major Depressive Disorder; Bipolar Disorder; Schizophrenia
Keywords: inpatients
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Schizophrenia | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: Feasibility Randomized Controlled Trial (RCT)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (HIIT) (Experimental): 50% of participants (inpatients with a diagnosis of severe mental illness) will be randomised to HIIT. HIIT will be conducted twice a week for 12 weeks using a stationary bike. Each session will have the following structure: 4-minute warm-up, followed by 5X1 minute intervals at 85-95% of maximum heart rate, interspersed with active pauses of 90 seconds cycling at approximately 60-70% of maximum heart rate, and a 4-minute cool-down. Each exercise session will take 19 minutes to complete (11 minutes of HIIT + warm-up and cool-down). However, the amount of HIIT will be adapted for people who may be unable to complete the above target and gradually build up until they can complete the recommended amount.
  All exercise sessions will be conducted in a 1:1 environment with a participant and a member of the research team who will supervise the exercise session.
  Interventions: Other: High Intensity Interval Training (HIIT)
- Treatment As Usual (TAU) (No Intervention): 50% of participants will be randomised to TAU. They will be provided with details of the local hospital gym availability and instructed to maintain their usual dietary habits

INTERVENTIONS:
Other: High Intensity Interval Training (HIIT) — HIIT is a type of exercise involving alternating short bursts of high intensity exercise with recovery periods of rest or light exercise.
  Arms: High Intensity Interval Training (HIIT)

SUMMARY:
People experiencing severe mental illnesses (SMI), including schizophrenia, psychosis, bipolar disorder and major depressive disorder, are prone to poorer physical health and increased incidences of premature mortality when compared to the general population (De Hert et al., 2009; Hert et al., 2011; Hennekens et al., 2005; Tiihonen et al., 2009 . High-intensity-interval-training (HIIT) is a type of exercise involving alternating short bursts of high intensity exercise with recovery periods of rest/ light exercise (Weston, Wisløff & Coombes, 2014). HIIT improves physical health, quality of life and cognition in the general population and in those with physical health disorders (Gomes-Neto et al., 2017; Hwang, Wu & Chou, 2011; Wen et al., 2019). It has been proposed that HIIT may improve symptoms, physical health and time to discharge among inpatients with SMI.

The research will involve three stages: 1) Focus groups, 2) A pilot study, 3) Follow-up qualitative interviews and focus groups.

Firstly, a series of focus groups with inpatients with SMI, carers of individuals with SMI and clinical staff will be conducted. The focus groups will scope perceptions of attitudes, and practicalities of a pilot RCT. The information gained will be used to inform a pilot HIIT trial which will evaluate whether HIIT is acceptable and feasible amongst this population group. Each focus group will run for ≈2 hours and will involve an open discussion about the benefits and barriers of conducting HIIT exercise sessions in a population with SMI.

Secondly, the HIIT pilot study will be trialed. The final protocol will be developed with feedback from the focus group but will involve an RCT where 12 weeks of HIIT will be compared to 12 weeks of treatment-as-usual (TAU). HIIT will be conducted, twice a week, in a supervised environment using a stationary bike. Inpatients with a diagnosis of SMI will be eligible to participate. Thirdly, follow-up qualitative interviews, with pilot study participants, those that withdrew and those that did not want to take part, and focus groups with clinical staff will address the acceptability and feasibility of HIIT.

DETAILED DESCRIPTION:
Setting:

All three stages will take place in various South London and Maudsley Hospital NHS Trust (SLaM) Adult Mental Health settings affiliated with the Maudsley Hospital and the Bethlem Royal Hospital, and at the Institute of Psychiatry, Psychology and Neuroscience (IoPPN).

Stage One:

A series of focus groups with inpatients with a diagnosis of SMI, carers of people with a diagnosis of SMI and clinical staff will scope perceptions of attitudes, and practicalities of a pilot RCT. It is expected that between 6-8 people will attend each focus group.

Up to 5 focus groups will be conducted, lasting two hours each, addressed at the following populations: 1) Clinical staff affiliated with SLaM; 2) Inpatients with a diagnosis of SMI who reside at the Maudsley Hospital and the Bethlem Royal Hospital, and their carers; 3) Carers recruited via the national carers' forum, a carers group in SLaM.

Procedure: A series of simple open-ended questions will be asked, and participants will answer verbally. The questions will address factors relevant to the pilot study design including optimal duration and intensity of exercise sessions; location of exercise sessions; procedures surrounding storage of exercise equipment; and procedure surrounding outcome assessments. An audio-recording will record responses to these questions when permission has been granted. The qualitative data gained from the questions asked as part of the focus group will be analysed using thematic analysis to understand the main themes.

Stage Two:

Part a- A pilot RCT will be conducted whereby inpatients with a diagnosis of SMI will be randomly allocated to either 12 weeks of HIIT or 12 weeks of TAU. For patients in the HIIT arm, HIIT will be conducted twice a week for 12 weeks using a stationary bike. Each session will have the following structure: 4-minute warm-up, followed by 5X1 minute intervals at 85-95% of maximum heart rate, interspersed with active pauses of 90 seconds cycling at approximately 60-70% of maximum heart rate, and a 4-minute cool-down. Assessment measures including a neuropsychological test battery; fitness test; and physical health checks will be conducted at baseline, 6-, and 12-weeks. Twenty inpatients will be recruited to each arm of the RCT (40 inpatients in total). This number is based on recruiting a big-enough sample to assess the feasibility of the study and on the resources available (Leon, Davis & Kraemer, 2011).

Pre-post intervention changes in will be measured, including changes in neuropsychological outcomes, fitness, physical health, and cardiovascular risk. A between-group analysis will also be conducted to see whether any changes in outcome differ from the control (TAU) group.

Part b- The RCT commenced in January 2020 using the above RCT procedure. Recruitment was halted in March 2020 at the start of the Covid-19 pandemic and HIIT sessions were ceased. The data gained will be analysed as above using an intention-to-treat basis.

In light of easing of lockdown the HIIT trial will resume using a remote cohort design. All eligible participants will receive HIIT, no randomisation will take place. A cohort design will be employed due to the smaller number of SMI patients receiving inpatient treatment during the outbreak/ slow resumption of inpatient admissions, thus it is unlikely that there will be enough numbers to randomise patients. The study primary and secondary outcomes remain the same.

HIIT sessions will resume remotely. This data will be analysed separately to existing data gathered from the RCT. A pre-post analysis on an ITT basis and a subgroup of those with 64% adherence will take place. The research team will conduct HIIT sessions remotely via a projector screen but a member of the ward will supervise sessions in person. Adverse events/ injuries/ difficulties will be observed by both the researcher remotely and the in-person staff member. Baseline and follow-up assessments will be conducted remotely via a projector screen/ telephone call for questionnaire measures.

A target of 6-8 patients will be recruited to the cohort study design.

Stage Three:

1. Qualitative interviews:

   Participants who completed the pilot study will be invited to take part in individual semi-structured follow-up qualitative interviews. Feedback regarding the acceptability and feasibility of the study will be sought. Additionally, feedback will be sought from those that withdrew from the study and those that did not agree to take part. The interviews will assess 1) how participants experienced the intervention, 2) if there are any parts of the intervention that could be improved, and what factors influenced people in completing/not completing the intervention. Interviews will take place on a one-to-one basis with a member of the research team and a participant. Each qualitative interview will be conducted within 3 weeks of each participant finishing the HIIT pilot study/ within 3 weeks of drop-out if time commitments permit. Responses will be recorded when permission has been granted. Overall, each individual interview will take 30- 60 minutes and will not require participants to participate in any follow-up tasks. The qualitative data gained from these questions will be analysed using thematic analysis to understand the main themes.
2. Focus groups:

Up to two focus groups with clinical staff at SLaM will be conducted and feedback regarding the acceptability and feasibility of the pilot HIIT study conducted in stage two of the research project will be sought. It is expected that between 6-8 people will attend each focus group. A series of simple open-ended questions will be asked, and participants will answer verbally. The questions will address staff's opinions regarding the acceptability and feasibility of conducting HIIT in a mental health setting. An audio-recording will record responses to these questions when permission has been granted. The qualitative data gained from these questions will be analysed using thematic analysis to understand the main themes. Overall, each focus group should take no more than 2 hours and will not require participants to participate in any follow-up tasks.

ELIGIBILITY:
Inclusion Criteria:

Stage 1 (Focus Groups):

* Capacity to provide informed consent.
* Aged ≥18 years.
* Either be: 1) Inpatients at SLaM with a diagnosis of SMI (Major Depressive Disorder, Bipolar disorder, Schizophrenia Spectrum Disorders, 2) Carers providing unpaid support to someone with a SMI, 3) Clinical staff at SLaM.

Stage 2 (HIIT Pilot RCT):

* Inpatients at SLaM with a diagnosis of SMI.
* Capacity to provide informed consent.
* Aged 18 -60.
* Ready to exercise according to the Physical Activity Readiness Questionnaire.

Stage 3 (Follow-up): Qualitative interview:

* inpatients who were eligible for stage 2.

Stage 3 (Follow-up): Focus group:

* staff who participated in stage 1.

Exclusion Criteria:

Stage 1 (Focus Groups):

* Is aged <18 years old.

Stage 2 (HIIT Pilot RCT) & Stage 3 qualitative interviews:

* Is aged <18 years old or >60 years old.
* Is pregnant.
* Has an eating disorder.
* Has a medical condition that impedes exercise, (as assessed via discussion with the patient's clinical team).

Stage 3 focus group:

* Did not complete stage one.

ALL STAGES:

* Is unable to provide informed consent.
* Is unable to understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-08-30 (Actual)

PRIMARY OUTCOMES:
Number of wards that agree to hosting the HIIT Pilot Study and number that do not agree to hosting the HIIT pilot study | Through study completion, an average of 1 year
  as assessed via a tally of acceptances and refusals
Number of people who consent to take part | Through study completion, an average of 1 year
  as assessed via a tally of acceptances and refusals
Average adherence to HIIT sessions and assessments | Throughout length of participation in the HIIT trial, 12 weeks
  as assessed via a record of number of HIIT sessions and number of assessments attended, and number of HIIT sessions and assessments not attended
Number of Participants With Treatment-Related Adverse Events | Through study completion, an average of 1 year
  as assessed via a tally of all medical effects observed and all medical effects reported by participants

SECONDARY OUTCOMES:
BMI | baseline, 6-weeks, 12-weeks
  BMI will be measured according to criteria set out by the International Diabetes Federation (IDF). A BMI between 18.5 to 24.9 will be interpreted as a healthy weight. Scores between 25 and 29.9 will be interpreted as overweight and a BMI >30kg/m² will be classified as central obesity.
Weight | baseline, 6-weeks, 12-weeks
  Weight will be measured in Kg using household scales. The investigators will assess whether weight decreases after participation in the HIIT trial.
Waist Circumference (WC) | baseline, 6-weeks, 12-weeks
  WC will be measured according to criteria set out by the International Diabetes Febderation (IDF). For Europids, a WC ≥ 94 cm and ≥ 80 cm indicates central obesity for men and women respectively. For persons from South Asia, China and Japan the cut-offs are ≥ 90 cm and ≥ 80 cm for men and women respectively.
Systolic and diastolic blood pressure | baseline, 6-weeks, 12-weeks
  Blood pressure will be measured using a blood pressure monitor. Higher systolic and diastolic blood pressure indicates lower cardiovascular function.
Maximal oxygen uptake (VO2max) | baseline, 6-weeks, 12-weeks
  VO2max will be measured using the YMCA cycle ergometer test which is a graded exercise test. Higher VO2max scores indicate greater cardiorespiratory fitness.
Gait speed | baseline, 6-weeks, 12-weeks
  The investigators will measure time taken to walk 6 meters. Longer times indicate reduced physical fitness.
Change in Montreal Cognitive Assessment (MoCA) score | baseline, 6-weeks, 12-weeks
  MoCA scores range between 0 and 30. Lower scores indicate worse cognitive functioning. A score of 26 or over is considered to be normal.
Change in global assessment of functioning scale (GAF) score | baseline, 6-weeks, 12-weeks
  GAF scores range from 0-100. Lower scores indicate worse global functioning. A score under 50 indicates severe impairment to functioning.
Change in Brief Psychiatric Rating Scale (BPRS) score | baseline, 6-weeks, 12-weeks
  The BPRS measures depression, anxiety, hallucinations and unusual behaviour. 24 items are rated from 1-7. A higher score indicates more severe psychiatric symptoms.
Change in the brief insomnia severity index (ISI) | baseline, 6-weeks, 12-weeks
  ISI scores range from 0-28. 0-7 indicates no clinically significant insomnia, 8-14 indicates sub-threshold insomnia and 15-28 indicates clinical insomnia.
Cigarette intake | baseline, 6-weeks, 12-weeks
  Participants will be asked how many cigarettes they smoke on a typical day.
Change in Depression Anxiety Stress Scale short version (DASS21) score | baseline, before and after the first HIIT session (or before and after 19 minutes of rest for the TAU arm), 6-weeks, 12-weeks
  The DASS21 contains 7 items for depression, 7 for anxiety and 7 for stress. Each subscale is scored from 0-42. Higher scores indicate higher levels of depression, anxiety and stress. Scores of 21, 15 and 26 indicate severe depression, anxiety and stress respectively.
Change in the Rosenberg Self-Esteem Scale (RSES) score | baseline, 6-weeks, 12-weeks
  RSES scores range from 0-30. Lower scores indicate lower self-esteem. A score under 15 may indicate problematic low self-esteem.
Change in the International Physical Activity Questionnaire (IPAQ) score | baseline, 6-weeks, 12-weeks
  Participants are asked to quantify how much physical activity they have completed over the past 7 days.
Change in the Behavioural Regulation in Exercise Questionnaire-3 (BREQ-3) score | baseline, 6-weeks, 12-weeks
  The BREQ contains 24 items with a score ranging from 0-4 for each item. The items are grouped into 6 factors with 4 items in each factor. Scores from each factor are combined using a weighting approach. Higher, positive scores indicate greater relative autonomy; lower, negative scores indicate more controlled regulation.
Change in the Short Warwick Edinburgh Mental Well-being Scale (WEMWBS) score | baseline, 6-weeks, 12-weeks
  Scores range from 7 to 35 and higher scores indicate higher positive mental well-being.

OTHER OUTCOMES:
Appetite cravings | before and after the first HIIT session (or before and after 19 minutes of rest for the TAU arm
  Participants will be asked: 'On a scale of 0-10 how much do you feel like smoking?' (0 will indicate no craving and 10 will indicate a craving)
Cigarette cravings | before and after the first HIIT session (or before and after 19 minutes of rest for the TAU arm
  Participants will be asked: 'On a scale of 0-10 how much do you feel like eating a snack right now? And if you do feel like eating what would it be?' (0 will indicate no craving and 10 will indicate a craving)
Change in Subjective Exercise Experiences Scale (SEES) score | before and after the first HIIT session (or before and after 19 minutes of rest for the TAU arm
  This questionnaire contains 12-items subdivided into three subscales to assess immediate feelings of positive well-being, psychological distress and fatigue. Each subscale contains the scores from 4-items rated on a 7-point Likert scale. Higher scores for each subscale indicated higher perceptions of positive well-being, psychological distress and fatigue respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Brendon Stubbs, Principal Investigator — King's College London
Locations (2):
- United Kingdom (2):
  - Bethlem Royal Hospital, South London and maudsley NHS Trust, London
  - Maudsley Hospital, South London and Maudsley NHS Trust, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leon AC, Davis LL, Kraemer HC. The role and interpretation of pilot studies in clinical research. J Psychiatr Res. 2011 May;45(5):626-9. doi: 10.1016/j.jpsychires.2010.10.008. Epub 2010 Oct 28. PMID 21035130
- [Background] DE Hert M, Correll CU, Bobes J, Cetkovich-Bakmas M, Cohen D, Asai I, Detraux J, Gautam S, Moller HJ, Ndetei DM, Newcomer JW, Uwakwe R, Leucht S. Physical illness in patients with severe mental disorders. I. Prevalence, impact of medications and disparities in health care. World Psychiatry. 2011 Feb;10(1):52-77. doi: 10.1002/j.2051-5545.2011.tb00014.x. PMID 21379357
- [Background] De Hert M, Dekker JM, Wood D, Kahl KG, Holt RI, Moller HJ. Cardiovascular disease and diabetes in people with severe mental illness position statement from the European Psychiatric Association (EPA), supported by the European Association for the Study of Diabetes (EASD) and the European Society of Cardiology (ESC). Eur Psychiatry. 2009 Sep;24(6):412-24. doi: 10.1016/j.eurpsy.2009.01.005. Epub 2009 Aug 13. PMID 19682863
- [Background] Hennekens CH, Hennekens AR, Hollar D, Casey DE. Schizophrenia and increased risks of cardiovascular disease. Am Heart J. 2005 Dec;150(6):1115-21. doi: 10.1016/j.ahj.2005.02.007. PMID 16338246
- [Background] Tiihonen J, Lonnqvist J, Wahlbeck K, Klaukka T, Niskanen L, Tanskanen A, Haukka J. 11-year follow-up of mortality in patients with schizophrenia: a population-based cohort study (FIN11 study). Lancet. 2009 Aug 22;374(9690):620-7. doi: 10.1016/S0140-6736(09)60742-X. PMID 19595447
- [Background] Weston KS, Wisloff U, Coombes JS. High-intensity interval training in patients with lifestyle-induced cardiometabolic disease: a systematic review and meta-analysis. Br J Sports Med. 2014 Aug;48(16):1227-34. doi: 10.1136/bjsports-2013-092576. Epub 2013 Oct 21. PMID 24144531
- [Derived] Martland R, Onwumere J, Stubbs B, Gaughran F. Study protocol for a pilot high-intensity interval training intervention in inpatient mental health settings: a two-part study using a randomised controlled trial and naturalistic study design. Pilot Feasibility Stud. 2021 Nov 8;7(1):198. doi: 10.1186/s40814-021-00937-6. PMID 34749822